CLINICAL TRIAL: NCT06988189
Title: Unmasking Concealed Arrhythmia Syndromes
Acronym: UCAS
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: REC 24/NS/0032
Record Dates: First submitted 2025-05-08; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Brugada ECG Patterns; Brugada Syndrome (BrS)
Keywords: Brugada syndrome; Ambulatory ECG; Wearable ECG; Long term continuous monitoring; AI ECG
MeSH Terms: conditions — Brugada Syndrome | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy volunteers: Volunteer participants with no cardiac structural or arrhythmic conditions.
  Interventions: Diagnostic Test: 12-lead ECG; Diagnostic Test: Continuous long term ambulatory ECG monitoring; Diagnostic Test: Ultra-high-frequency ECG
- Manifest Arrhythmia Syndrome: Manifest arrhythmia syndrome patients (patients with an arrhythmic syndrome with an abnormal ECG)
  Interventions: Diagnostic Test: 12-lead ECG; Diagnostic Test: Continuous long term ambulatory ECG monitoring; Diagnostic Test: Ultra-high-frequency ECG
- Concealed Arrhythmia Syndrome: Concealed arrhythmia syndrome patients (patients with a normal ECG with a known underlying arrhythmic diagnosis)
  Interventions: Diagnostic Test: 12-lead ECG; Diagnostic Test: Continuous long term ambulatory ECG monitoring; Diagnostic Test: Ultra-high-frequency ECG

INTERVENTIONS:
Diagnostic Test: 12-lead ECG — 12-lead ECG from a conventional ECG machine
Diagnostic Test: Continuous long term ambulatory ECG monitoring — Continuous long term ambulatory ECG monitoring using wearable ECG or cardiac monitor
Diagnostic Test: Ultra-high-frequency ECG — Ultra-high-frequency ECG acquired using specific acquisition equipment

SUMMARY:
This study seeks to evaluate whether using non-invasive electrocardiograph (ECG) techniques, including long term ECG monitoring with wearable ECGs, can improve the detection of concealed Brugada syndrome.

DETAILED DESCRIPTION:
Application of long term continuous ECG monitoring via ECG wearables and ambulatory ECG monitors to detect manifestations of Brugada syndrome. This approach will be combined with development of an AI (artificial intelligence) enabled ECG platform to automate Brugada ECG detection and analysis.

The protocol will comprise the following parts:

Study A: Brugada ECG AI development. This will automate the recognition of the type 1 Brugada ECG pattern on 12 lead ECGs.

Study B: Remote arrhythmia diagnostics. A prospective observational study whereby recruited participants will be fitted with a wearable ECG or cardiac monitor to undergo continuous long term ambulatory ECG monitoring. The algorithms developed in study A will be applied to long term ECG data captured in this study.

Study C: Arrhythmic risk stratification using ultra-high-frequency ECG. This exploratory study will look for markers of arrhythmic risk in patients with manifest and concealed arrhythmia syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Adults willing to take part
* Able to give consent

Exclusion Criteria:

* Unable to give consent
* Children age < 18 years and adults > 100 years old

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteer controls, patients with a diagnosis of Brugada syndrome, patients with a diagnosis of idiopathic VF syndrome and patients with other inherited arrhythmogenic conditions.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, and area under the curve (AUC) of AI algorithm for detection of Brugada type 1 ECG pattern on 12-lead ECGs. | At completion of algorithm validation, approximately 12 months after study start
  Assessment of performance and accuracy of AI ECG detection algorithm for type 1 Brugada ECG.
Detection rate of Brugada ECG pattern using extended-duration multi-electrode ambulatory ECG monitoring (wearable ECG) in patients with concealed Brugada syndrome. | Up to 12 months from enrolment
  AI ECG detection algorithm, developed in Study A, applied to full ECG recording to detect Type 1 Brugada ECG pattern.
Number of cases of Brugada or Long QT Syndrome (LQTS) detected using extended-duration multi-electrode ambulatory ECG monitoring in patients with idiopathic ventricular fibrillation (VF), after application of AI ECG detection algorithms. | Up to 12 months from enrolment
  AI ECG detection algorithms applied to full ECG recording to detect Type 1 Brugada ECG pattern or LQTS unmasking.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Whinnett, PhD, Study Chair — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gray B, Kirby A, Kabunga P, Freedman SB, Yeates L, Kanthan A, Medi C, Keech A, Semsarian C, Sy RW. Twelve-lead ambulatory electrocardiographic monitoring in Brugada syndrome: Potential diagnostic and prognostic implications. Heart Rhythm. 2017 Jun;14(6):866-874. doi: 10.1016/j.hrthm.2017.02.026. PMID 28528724

DOCUMENTS (2):
  • Study Protocol (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT06988189/Prot_000.pdf
  • Informed Consent Form (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT06988189/ICF_001.pdf